CLINICAL TRIAL: NCT06593925
Title: Assessment of Polyoxymethylene (POM) as a Material for the Outer Crowns and Telescopic Denture's Framework in the Treatment of Subtotal Edentulism
Brief Title: Polyoxymethylene (POM) in the Production of Telescopic Denture in Older Adults With Subtotal Edentulism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Djurdja Nedeljkovic, PhD student, University of Belgrade
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No 36/29; 19-11-2021
Record Dates: First submitted 2024-07-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Subtotal Edentulism
Keywords: polyoxymethylene; double crowns; telescopic denture; conventional complex partial denture with clasps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Polyoxymethylene telescopic denture (Experimental)
  Interventions: Device: Production of polyoxymethylene telescopic denture
- Conventional complex partial denture with clasps (Active Comparator)
  Interventions: Device: Production of conventional complex partial denture with clasps

INTERVENTIONS:
Device: Production of polyoxymethylene telescopic denture — Remaining teeth will be prepared by conventional grinding technique, followed by impression, casting and scanning with extra oral scanner. Inner telescopic crowns will be made of cobalt-chromium alloy by milling technique and outer crowns together with denture framework will be made of polyoxymethylene by the method of single phase injection moulding. Denture delivery is done by inserting both inner and outer crown at the same time, during which the inner crown is cemented to the abutment tooth and the contact surfaces of the outer and inner crown are isolated so that the outer crown and denture framework can be removed.
  Arms: Polyoxymethylene telescopic denture
Device: Production of conventional complex partial denture with clasps — A conventional complex partial denture is a removable partial denture with clasps combined with metal-ceramic surveyed crowns with milled surfaces for removable dentures. The metal-ceramic surveyed crowns are shaped in such a way that they build a morphological and functional whole with complementary elements of the removable partial denture's framework. In the control group, as well as in the experimental group, the remaining teeth are prepared using a conventional grinding technique, then an impression is taken for dedicated metal-ceramic crowns, casting, and milling of crowns, ceramic sintering, impression through the metal-ceramic surveyed crowns and fabrication of a removable partial denture's framework with clasps using the casting method. Dedicated fixed restorations will be made of Co-Cr alloy inside the crown and ceramic layer on the surface, and the framework and clasps of the removable partial denture will be made of Co-Cr-Mo alloy.
  Arms: Conventional complex partial denture with clasps

SUMMARY:
The mail goal of this study is to evaluate the success of the prosthetic treatment with telescopic removable partial denture with framework made of polyoxymethylene (POM). In accordance with the growing older population, who often require complex dental care, it is very important to test simple yet effective and safe solutions. Bearing in mind that POM has proven to be a good solution for conventional removable partial dentures with clasps (RPD), and that it is quite common to have 2-3 remaining teeth, a denture with a framework made of light and flexible material such as POM present a good solution. The hypothesis is that a POM telescopic denture is clinically as adequate, effective and safe as the conventional complex cobalt chromium molybdenum alloy denture with clasps. Telescopic denture should provide better comfort and longevity compared to conventional RPD because of axial loading of the abutment teeth and no negative biological effect of clasps. Moreover, conventional telescopic denture is made of precious alloys which increase their cost; therefore, POM telescopic denture present great advantage in cost/effective treatment. Telescopic crowns are comprised of inner and outer crowns; accordingly, telescopic denture represent a type of complex denture where one part is fixed on the remaining teeth (inner crowns) and other part (outer crowns and denture framework) is removable.

The key factors that will define the success of the treatment will be: assessment of dentures' retention, oral health related quality of life, presence of biological complications, presence of mechanical complications, denture appearance and chewing function assessment.

DETAILED DESCRIPTION:
The study is designed as experimental research, therefore it is necessary to have an experimental and a control group. The experimental group would consist of patients who will be prosthetically rehabilitated with telescopic dentures made of polyoxymethylene, and the control group would consist of patients with a conventional complex removable partial denture with metal alloy clasps. The study will be conducted at the Clinic for Prosthodontics, Faculty of Dentistry, University of Belgrade. A patient who needs prosthetic rehabilitation and meets the criteria for inclusion in this study will be referred to the study chair, who based on the anamnesis, clinical examination, and analysis of the tomography, will decide whether the patient is suitable for the study. The principal investigator will inform the patient about the stages of production of prosthetic devices and the number of required visits. Also, the patient must sign an informed consent to participate in the study and read a detailed explanation about the type of prosthetic device that will be made for him. The principal investigator will randomly assign the selected patients to the experimental and control groups. The main stages of the protocol which will be done by principal investigator are: recruitment of patients, recording of data on detailed anamnesis and clinical examination, photographs of patients and dentures on the day of delivery and at control examinations, and analysis of all obtained results. The clinical phases of the research will be performed by different clinicians, but always the same for the same patient. All phases of the research will be under the supervision of the study chair. In addition to demographic data, it is necessary to obtain information about: the patients' health condition, allergies, undergoing radio/chemo therapy (before/at the time of arrival/planned in the future), smoking status, the presence of bad habits and the existence of prosthetic devices in the past (type of prosthetic devices and how long it was worn).

The clinical examination is planned to obtain information about the patients' skeletal class, the number, arrangement, and condition of the remaining teeth, the number of functional units of the teeth, the presence of mucogingival anomalies/ exostoses/ tuber hypertrophy/ gothic palate/ mobile alveolar ridge and the type of tooth replacement in the antagonistic jaw (if the same exists). The clinical phases of the research will include the process of production of dentures, notation of mechanical complications, assessment of retention force by the patient and clinician, filling in the GOHAI questionnaire, determination of the CPITN index, assessment of the appearance of the dentures, and assessment of chewing efficiency (two-color chewing gum test) and chewing ability (CFQ questionnaire). All parameters will be recorded on the day of delivery and at control examinations after 6 months and after a year, except CFQ questionnaire and two-color chewing gum test which will be measured only after on year of use, after complete adaptation of new dentures is achieved.

Mechanical complications will include: a fracture of the denture's base, artificial tooth falling out of the denture, disconnection between POM framework and artificial teeth, and fracture of the outer telescopic crown. The outcome of therapy will be better if fewer mechanical complications occur. Biological complications occur if the prosthetic device disturbs the periodontal tissue and/or teeth. Biological complications will be assessed by the CPITN index (Community Periodontal Index of Treatment Needs) and recording the need for endodontic treatment or extraction of retention teeth. CPITN index will be used due to its simplicity of execution, reliability, objectivity, and reproducibility. Identification of the condition of periodontal tissues will be done based on inspection and periodontal probing of the teeth from all four sides of the teeth, based on which values from 0-5 will be assigned (0=healthy gingiva and periodontal tissues, 1=bleeding on provocation by probing with a periodontal probe, 2=existence of supragingival calculus, 3=existence of periodontal pockets, 4=existence of periodontal pockets deeper than 6mm, 5=missing tooth due to extraction or tooth is indicated for extraction). The outcome of therapy will be better if the value of the CPITN index is the same or lower at control examinations than at the time of delivery and if the values of the CPITN index are the same or lower in the experimental group than in the control group. Also, the outcome of therapy will considered better if at the time of the control examination, there is no need for tooth extraction or endodontic treatment of retention teeth. The appearance of the denture will be assessed based on the presence of pigmentation and/or fissures. The appearance of the dentures will be assessed by analyzing photos of the denture parts, taken with the same camera, in daylight, and on the same surface. Photographs will be taken of the major connector and parts of the framework around each retention tooth. Appearance scores will range from 0-6 (0=no pigmentation and fissures, 1=presence of moderate pigmentation without fissures, 2=presence of marked pigmentation without fissures, 3=presence of moderate pigmentation with one fissure, 4=presence of moderate pigmentation with multiple fissures, 5=presence of marked pigmentation with one fissure, 6=presence of marked pigmentation with multiple fissures). The outcome of therapy will be better if the appearance scores of the dentures are lower during follow-up examinations compared to the day of delivery. The assessment of the retention force of the dentures will be done by the assessment of the patient and the clinician (always the same for each patient) by grading on a Likert scale (1-10). The assessment will be done manually when the denture is removed. A better result of therapy is to keep the same point on the Likert scale or to assign a better point compared to the day of delivery. The patients' quality of life related to oral health will be assessed subjectively using the GOHAI (Geriatric Oral Health Assessment Index) questionnaire. This questionnaire will be used because of its sensitivity, specificity, and positive predictive value. This questionnaire was developed as an indicator of self-perception of dental problems in the older population. Although it was originally developed in English, a cultural and linguistic adaptation of the questionnaire was carried out in Serbian. The questionnaire is composed of 12 questions, nine of them are formulated in a negative and three in a positive form. A copy of the questionnaire will be given to patients to enable them to read the questions themselves, and if reading or understanding is difficult, the clinician will ask questions and provide explanations without suggesting a potential answer. Patients will answer questions using a Likert scale (1-5) and rate how often the problem has been present/absent in the last three months. There are five answer categories for each question (1=always, 2=often, 3=sometimes, 4=rarely, 5=never). Results from positively worded questions will be reversed during statistical data processing so that the directions of all responses are the same. The overall score of the GOHAI questionnaire has a value of 60, which indicates a better patients' quality of life, while a score of 12 represents a markedly impaired patients' quality of life. The chewing function as an important indicator of quality of life will be evaluated subjectively and objectively. As an indicator of the subjective evaluation of the chewing function (chewing ability), the CFQ questionnaire (chewing function questionnaire) will be used, which is the first one-dimensional questionnaire related to the chewing function. The CFQ questionnaire contains 10 questions. Patients will answer questions using a Likert scale (0-4) and will assess how often they have a particular problem in the past 7 or 14 days. Zero indicates that they have no problems, and higher numbers indicate more serious problems, as well as the complete impossibility of consuming any of the listed foods (0=never, 1=rarely, 2=occasionally, 3=often, 4=very often). The total score of the CFQ questionnaire has a maximum value of 40, which indicates the greatest chewing difficulties, while a score of 0 represents the absence of the same. In order to objectively evaluate the chewing function (chewing efficiency), the two-color chewing gum test will be used. The samples will be Airwaves chewing gum, sugar-free, with sweetener, size 23x12x8mm. Two types were used: blue (menthol and eucalyptus flavor) and yellow (menthol and melon flavors), which are suitable for this type of research because in contact with saliva and under the action of the bite force, they don't change color and don't stick to dentures. This experiment is planned to last approximately 1 minute and it will mean 20 chewing cycles of a sample composed of 2 chewing gums (blue and yellow). The number of chewing cycles will be counted by the clinician. Each chewed sample will spit out into transparent plastic bags and then flattened to a thickness of 1 mm by pressing with a glass plate under manual pressure. Both sides of the sample will be photographed with a camera 16 Mpa, ISO-125, f/2.2, focal length 26mm. Each pair of photos will be converted into one photo, with a resolution of 300 dpi, which will be saved in .JPEG format. Such a photo will be entered into the commercially available computer program ViewGum, which was specially developed for colorimetric analysis of chewed samples. As the software shows the differences in the homogeneity of the samples numerically, the parameter of importance for examining the chewing efficiency is the Z-score. Lower Z-score values will mean that the patient chewed the given sample better.

All data collected during the study will be analyzed by the principal investigator, using the statistical software SPSS version 22. Absolute and relative numbers will be used for attributive features of observation, as methods of descriptive statistics, and for numerical features of observation, measures of central tendency and measures of dispersion will be used. Comparisons of the frequency of repetition of the analyzed attributive features of observation between groups will be performed using the Chi-square test and Fisher's exact test. The one-sample Kolmogorov-Smirnov test will be used to test the normality of the data distribution. Depending on the nature of the data distribution, an appropriate test (parametric or non-parametric) will be chosen for the analysis of the numerical features of the observation. To compare the obtained results between two groups, which behave according to the type of normal distribution, the parametric tests Student's T-Test (for unrelated samples) and T-test diff. (for related samples) will be used and for comparisons between three or more groups One-way ANOVA test (for unrelated samples) and one-factor analysis of variance (for related samples). Non-parametric tests will be used to analyze data that don't behave according to the type of normal distribution, whereby the Wilcoxon test (for related samples) and the Mann-Whitney U Test (for unrelated samples) will be used to analyze the results between two groups and to analyze the results between three or more groups, the Friedman test (for related samples) and the Kruskall-Wallis Test (for unrelated samples) will be used. Pearson's and Spearman's correlation coefficients will be used to determine the correlation between the measured parameters. The value p<0.05 will be used for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 and over
* patients with subtotal edentulism
* patients who sign an informed consent for participation in the study
* retention teeth must have a minimum crown/root ratio of 1:1
* retention teeth must have sufficient tooth substance (at least two walls)

Exclusion Criteria:

* patients younger than 65 years
* patients with temporomandibular joint dysfunction
* patiens with bruxism
* presence of intrabony defects around the retention teeth
* presence of pathological tooth mobility
* presence of periapical inflammatory processes, abscesses and fistulas in the region of retention teeth
* presence of fetor and suppuration from periodontal pockets of retention teeth

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with equal or greater prosthetic rehabilitation success treated with POM telescopic denture compared to conventional complex removable partial denture assessed by a success indicator | 1 year
  The success indicator are appearance of recording mechanical complications (presence and absence), biological complications (CPITN index with scale from 0-5 and recording the need for endodontic treatment or extraction of retention teeth), denture appearance (presence of pigmentation and/or fissures wih scale from 0-6), retention force assessment by patients and clinician (on a Likert scale from 1-10), GOHAI questionnaire (12 questions with Likert scale from 1-10, maximum scores of 60) and tests to assess the chewing ability-the CFQ questionnaire (10 questions with Likert scale from 0-4, maximum scores of 40) and chewing efficiency -the two-color chewing gum test (the parameter of importance is Z-score).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Popovac, Study Chair — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Denatal medicine, University of Belgrade, Belgrade, Serbia